CLINICAL TRIAL: NCT02803775
Title: Paced And Sensed Electrical Delay in CRT Therapy (PASED CRT)
Acronym: PASED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Heart and Lung Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2K15-03
Record Dates: First submitted 2016-06-07; First posted 2016-06-17 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Paced (Active Comparator): Paced arm in which the left heart lead electrode is selected utilizing the longest time to when patient right ventricle lead is pacing. The result of the pacing algorithm becomes the patient's pacing location for the study duration (self-assigned algorithm within this cohort).
  Interventions: Device: CRT Algorithm
- Sensed (Active Comparator): Sensed arm is based on the longest time that patient own heart's conduction reaches the left heart lead electrode.The result of the sensing algorithm becomes the patient's pacing location for the study duration (self-assigned algorithm within this cohort).
  Interventions: Device: CRT Algorithm

INTERVENTIONS:
Device: CRT Algorithm — Programming based on Electrogram measurement

SUMMARY:
Cardiac resynchronization therapy (CRT) is a well established clinical therapy for patients with symptomatic left ventricular systolic dysfunction and electrocardiographic QRS duration of 120 ms or greater. Multicenter trials have consistently demonstrated CRT "non responder" rates of 32-43% at 6 months. Subsequent studies have shown that utilizing echocardiographic-guided device reprogramming for optimal atrio-ventricular (A-V) and interventricular (VV) delays at rest have improved clinical response. Recently, an echocardiographically validated automated pacemaker programmer-based intra-cardiac electrogram (IEGM) algorithm has been developed for rapid optimization of sino-ventricular (P-V), A-V and V-V delays at resting heart rates that is partially based on the interventricular conduction time delays. Nevertheless, controversy still persists as to the applicability of both echocardiographic and IEGM derived algorithms at elevated heart rates, as with physical activity, when patients are more likely to experience symptoms related to poor cardiac output.

Recent studies have shown clinical benefits of pacing from sites of late intrinsic activation or intra-ventricular conduction delays (IVCD). Some studies have utilized the intrinsic SENSED IVCD method while others used the right ventricle (RV)-PACED IVCD. There have not been any studies to date that compare both methods to determine if one may yield a better clinical outcome with lower non-responder rates.

This study predicts that the RV paced IVCD method will provide better clinical outcomes than the longest RV sensed IVCD as determined by the clinical composite score.

The study is a prospective double blind study with an additional cross-over group consisting only of non-responders to compare the clinical response in 72 patients receiving CRT therapy. After successful CRT-D implantation and before hospital discharge patients will be randomly assigned in a 1:1 fashion to Group 1 (SENSED) or Group 2 (PACED). The patient will complete a Minnesota Living with Heart Failure questionnaire, compare echocardiographic data and be assessed by a blinded nurse and physician prior to discharge and at each follow up visit to maintain the double blind design.

After 3 months of follow-up, non-responders from each group will be crossed-over to the other group and followed for an additional 3 months. Clinical data will be collected at the end of that 3 months and compared looking at changes in symptoms, ejection fraction (EF) and other echocardiographic measurements, New York Heart Assocation Function Class ( NYHA) class, clinical composite scores (CCC), device interrogation data and hospital admissions between the two groups to see if there is a statistical difference.

ELIGIBILITY:
Inclusion Criteria:

* Ejection Fraction less than or equal to 35%
* American College of Cardiology (ACC)/American Heart Association (AHA) indicated patients with surface ECG QRS duration greater than or equal to 120ms

Exclusion Criteria:

* Previously placed left ventricular (LV) lead receiving CRT therapy for greater than 3 months
* Pregnant or planning to become pregnant
* Classification of status 1 for cardiac transplant patients for next 9 months,
* Participating in another clinical investigation with an active treatment arm
* Life expectancy of less than nine months
* Age less than 18 years
* Inability to successfully implant LV lead
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Change in six-minute walk distance | Baseline, 3 months and 6 months. The six month assessment is optional for non-responders participating in crossover option
  Six-minute walk distance (measured in meters)

SECONDARY OUTCOMES:
Clinical Composite Score | Baseline, 3 months and 6 months. The six month assessment is optional for non-responders participating in crossover option
  Packer Clinical Composite Score Questionnaire captures the following outcomes: death (yes/no field), hospitalizations (yes/no field), global patient assessment (likert scale 1-5 points) , functional heart class (I, II, III, IV).

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Corbisiero, MD, Principal Investigator — Deborah Heart and Lung Center; Pedram Kazemian, MD, Principal Investigator — Deborah Heart and Lung Center
Locations (1):
- Deborah Heart and Lung Center, Browns Mills, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Packer M. Proposal for a new clinical end point to evaluate the efficacy of drugs and devices in the treatment of chronic heart failure. J Card Fail. 2001 Jun;7(2):176-82. doi: 10.1054/jcaf.2001.25652. PMID 11420770